CLINICAL TRIAL: NCT02534402
Title: Clinical Implementation and Outcomes Evaluation of Blood-Based Biomarkers for COPD Management: COPD Prednisone Sub-Study
Brief Title: Prednisone Administration in Quiescent COPD Patients to Determine the Effect on Gene Expression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Don Sin, Dr. Don Sin, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H15-01147
Record Dates: First submitted 2015-08-26; First posted 2015-08-27 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Biomarkers; Genomics; Prednisone
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisone Group (Experimental): 30mg of prednisone PO (orally) everyday for 5 days.
  Interventions: Drug: Prednisone
- Control Group (No Intervention): no treatment

INTERVENTIONS:
Drug: Prednisone — Administration of prednisone to determine the effect on whole blood gene expression.
  Other Names: Deltasone; Orasone; Prednicen-M; Liquid Pred
  Arms: Prednisone Group

SUMMARY:
In this study, prednisone dose, day/time administration will be controlled in a stable COPD patient population to determine its effect on peripheral whole blood gene expression. This data has never been collected in a COPD population using the investigators' chosen platform for gene expression (Affymetrix Human Gene 1.1 ST). Conducting this experiment is essential for achieving the broader aims of an already existing and related study titled "Clinical Implementation and Outcomes Evaluation of Blood-Based Biomarkers for COPD Management" study. As part of this existing study, blood is being collected from hospitalized and non-hospitalized COPD patients in order to develop a blood-based biomarker test for the diagnosis and prediction of acute exacerbation of COPD (AECOPD). The majority of these patients were administered prednisone as part of standard care for the treatment of AECOPD. As such, the effect of prednisone on gene expression needs to be ruled out.

DETAILED DESCRIPTION:
The course of COPD is frequently complicated by periods of exacerbation (worsening symptoms) related to infections, pollution, other diseases or poor management of disease. These periods result in urgent visits to physician offices or emergency rooms accounting for the leading cause of hospitalizations. In terms of patient care, physicians lack objective measurements to accurately risk-stratify patients and monitor the effectiveness of interventions provided for their patients. Regrettably, there are no blood tests that can predict who will and will not get AECOPD to require hospitalization. Additionally, current therapies for COPD are only modestly effective in reducing exacerbations. A major challenge in COPD drug development and patient care is the lack of markers, surrogate or otherwise, that can be used to predict outcomes such as hospitalization or mortality.

These critical barriers to drug development and improved patient care could be addressed by the development and clinical implementation of diagnostic and predictive AECOPD biomarkers. This is the aim of an already existing and related study titled "Clinical Implementation and Outcomes Evaluation of Blood-Based Biomarkers for COPD Management study". This study has been enrolling COPD patients since July 2012. The majority of the the study patients were on prednisone at the time of blood collection and at enrollment.

The analyses of publicly available datasets make it abundantly clear that prednisone has important and wide-ranging effects on peripheral whole blood gene expression. These data are insufficient, however, because they cannot inform disease specific effects on gene expression. In addition, because these studies were carried out using a different gene expression platform, they cannot be used to estimate the probeset-specific prednisone effects.

Therefore, the investigators need to ensure that the gene expression associated with AECOPD is not in fact a result of the drug effect. Conducting this study will help us answer this question.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with COPD

Exclusion Criteria:

* Participants currently taking prednisone
* Participants who received prednisone within the last 2 weeks
* Participants who were hospitalized in the last 2 weeks for COPD or a related respiratory condition

Ages: 19 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Effect of prednisone on peripheral whole blood gene expression | Period of 5 days
  Effect of prednisone on peripheral whole blood gene expression of stable COPD patients, assayed using Affymetrix Human Gene 1.1 ST microarrays. This outcome measure will be assessed at each blood draw.

CONTACTS AND LOCATIONS:
Overall Officials: Donald D Sin, MD, MPH, Principal Investigator — University of British Columbia, St. Paul's Hospital, James Hogg Research Centre
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Global Initiative for Chronic Obstructive Lung Disease, Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Pulmonary Disease (Updated 2009). http://www.goldcopd.com/Guidelineitem.asp?l1=2&l2=1&intId=2003.
- [Background] Chapman KR, Bourbeau J, Rance L. The burden of COPD in Canada: results from the Confronting COPD survey. Respir Med. 2003 Mar;97 Suppl C:S23-31. doi: 10.1016/s0954-6111(03)80022-7. PMID 12647940
- [Background] Mittmann N, Kuramoto L, Seung SJ, Haddon JM, Bradley-Kennedy C, Fitzgerald JM. The cost of moderate and severe COPD exacerbations to the Canadian healthcare system. Respir Med. 2008 Mar;102(3):413-21. doi: 10.1016/j.rmed.2007.10.010. Epub 2007 Dec 20. PMID 18086519
- [Background] Murray CJ, Lopez AD. Alternative projections of mortality and disability by cause 1990-2020: Global Burden of Disease Study. Lancet. 1997 May 24;349(9064):1498-504. doi: 10.1016/S0140-6736(96)07492-2. PMID 9167458
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Sin DD, McAlister FA, Man SF, Anthonisen NR. Contemporary management of chronic obstructive pulmonary disease: scientific review. JAMA. 2003 Nov 5;290(17):2301-12. doi: 10.1001/jama.290.17.2301. PMID 14600189
- [Background] Malhotra S, Man SF, Sin DD. Emerging drugs for the treatment of chronic obstructive pulmonary disease. Expert Opin Emerg Drugs. 2006 May;11(2):275-91. doi: 10.1517/14728214.11.2.275. PMID 16634702
- [Background] Vestbo J, Anderson W, Coxson HO, Crim C, Dawber F, Edwards L, Hagan G, Knobil K, Lomas DA, MacNee W, Silverman EK, Tal-Singer R; ECLIPSE investigators. Evaluation of COPD Longitudinally to Identify Predictive Surrogate End-points (ECLIPSE). Eur Respir J. 2008 Apr;31(4):869-73. doi: 10.1183/09031936.00111707. Epub 2008 Jan 23. PMID 18216052
- [Background] Kuzyk MA, Smith D, Yang J, Cross TJ, Jackson AM, Hardie DB, Anderson NL, Borchers CH. Multiple reaction monitoring-based, multiplexed, absolute quantitation of 45 proteins in human plasma. Mol Cell Proteomics. 2009 Aug;8(8):1860-77. doi: 10.1074/mcp.M800540-MCP200. Epub 2009 May 1. PMID 19411661
- [Derived] Takiguchi H, Chen V, Obeidat M, Hollander Z, FitzGerald JM, McManus BM, Ng RT, Sin DD. Effect of short-term oral prednisone therapy on blood gene expression: a randomised controlled clinical trial. Respir Res. 2019 Aug 5;20(1):176. doi: 10.1186/s12931-019-1147-2. PMID 31382977